CLINICAL TRIAL: NCT06951607
Title: An Innovative Approach to the Management of Proximal Interphalangeal (PIP) Joint Injuries
Brief Title: Management of Proximal Interphalangeal (PIP) Joint Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-240
Record Dates: First submitted 2025-03-18; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Interphalangeal Joint Injury
Keywords: PIP Injury; Coban wrap; Neoprene Sleeve; Interphalangeal Joint

STUDY DESIGN:
Intervention Model Description: The study will take place at St. Joseph's Health Centre, Unity Health Toronto, in Toronto, Canada. The St. Joseph's site is capable of recruiting the required number of patients (40 total) for both the control (Group 1 - coban treatment) and the innovative treatment group (Group 2 - custom neoprene sleeve). The study design will be a randomized control trial, where participants will be randomly assigned to one of the two treatment groups, with 20 participants assigned to each treatment modality. Patients will be observed over a 6-month period, and outcome measures will be collected at initial assessment, 2 weeks, 4 weeks, 3 months and 6 months. Prior to study enrollment, written informed consent will be obtained from all participants.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coban wrap (Active Comparator): The Coban wrap is a compressive adhesive bandage used to joint injuries. Participants in this arm will receive a Coban wrap as a form of treatment with outcome measures occurring at the initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  Interventions: Other: Coban wrap
- Neoprene Sleeve (Experimental): Neoprene sleeve is an innovative treatment approach, it consists of a synthetic rubber-like material used to provide compressive support. Participants in this arm will receive a sleeve as a form of treatment with outcome measures occurring at the initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  Interventions: Other: Neoprene sleeve

INTERVENTIONS:
Other: Coban wrap — A Coban bandage or wrap is a self-adhering elastic wrap that sticks to itself but not to skin or clothing. It is commonly used as a wrap on limbs due to its ability to adhere to itself and not loosen. Coban is often used as a compression bandage
  Arms: Coban wrap
Other: Neoprene sleeve — Neoprene sleeve is an innovative treatment approach, it consists of a synthetic rubber-like material used to provide compressive support. Neoprene sleeves can provide protection, light compression and mild extension support while allowing full finger flexion.
  Arms: Neoprene Sleeve

SUMMARY:
This project seeks to compare the treatment efficacy of two different approaches to treating interphalangeal joint (PIP) joint injuries. The investigators will compare two participant groups undergoing treatment using the current treatment standard (Coban wrap) as well as an innovative treatment approach (neoprene sleeve) in treating the PIP joint injury.

DETAILED DESCRIPTION:
Hand injuries, specifically those involving the proximal interphalangeal joint (PIP) can be difficult to treat. These stubborn injuries leave patients with pain, edema, and limitation in function and changes in the aesthetics of the hand. This project would randomize patients with PIP joint injuries including dislocation, volar plate, intra-articular fracture and chip avulsion fracture with ligamentous injury into two groups. The first group will receive the usual treatment including active range motion, edema control - contrast bath and coban. The second group would receive similar treatment except a custom neoprene sleeve will be used in place coban. Outcome measures would include: Numeric Pain Rating Scale (NPRS), measure of patient satisfaction and compliance with the coban vs a custom neoprene sleeve and a measure of hand function (Patient Rated Wrist/Hand Evaluation) as well as a range of motion and edema.

ELIGIBILITY:
Inclusion criteria

* Read/write and speak/understand English
* Capable of understanding the various questionnaires that will be employed to collect outcome measures

Exclusion Criteria:

* Participants who do not meet all of the aforementioned criteria
* Participants with any injuries specific to the treatment finger, or if there is any underlying disease affecting the PIP joint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Edema | The outcome measures will be collected at various intervals, such as initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  The aim of the current study is to compare the treatment efficacy of a custom neoprene sleeve vs. a coban wrap in treating PIP joint injuries. In order to measure to measure treatment changes in edema (swelling) for PIP joint injuries. Edema will be measured using an instrument consisting of ring gage to determine whether the patient has experienced a decrease in swelling based on the circumferential numerical measurement comparison from their previous visit.
Changes in Pain | The outcome measures will be collected at various intervals, such as initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  The aim of the current study is to compare the treatment efficacy of a custom neoprene sleeve vs. a coban wrap in treating PIP joint injuries. The second primary outcome measure of interest is the level of pain that a patient may be experiencing at various intervals post injury, which can be measured using the Numeric Pain Rating Scale (NPRS).

SECONDARY OUTCOMES:
Range of Motion | The outcome measures will be collected at various intervals, such as initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  To measure range of motion during patient visit intervals, clinicians will be using an instrument known as a goniometer to determine the extent of which the patient has regained their range of motion post injury between the two treatment conditions (Coban wrap vs. neoprene sleeve).
Function and Appearance | The outcome measures will be collected at various intervals, such as initial visit, 2 weeks, 4 weeks, 3 months and 6 months.
  To measure function and appearance, clinicians will be administering the Patient Rated Wrist/Hand Evaluation (PRWHE) to determine the extent to which patients report regaining the function of their finger joints post injury, the scale includes a section which addresses patients' perceptions around appearance.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Ellis, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
The research will be published and disseminated within the organization and/or in a scientific journal.
Supporting Information: Study Protocol
Time Frame: After the data has been collected and analyzed.
Access Criteria: Only the study personnel have access to the study information.